CLINICAL TRIAL: NCT05863754
Title: Grasp-Release Assessment of a Networked Neuroprosthesis Device
Acronym: GRANND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Anne Bryden, Principal Investigator, MetroHealth Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB20-00854
Record Dates: First submitted 2023-04-28; First posted 2023-05-18 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury at C5-C7 Level; Spinal Cord Injuries; Spinal Cord Injury Cervical
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Experimental: Intervention - implant neuroprosthesis (Experimental): Receives implanted networked neuroprosthetic system for arm and hand function. Undergoes functional training and assessment.
  Interventions: Device: Networked Neuroprosthesis Device

INTERVENTIONS:
Device: Networked Neuroprosthesis Device — The Networked Neuroprosthesis Device is an implantable, configurable neuromodulation platform that provides functional movement by the coordinated activation of peripheral neural pathways activating innervated paralyzed muscles, and sensing of physiological signals.

SUMMARY:
The overall objective of this trial is to characterize the safety and effectiveness of the Networked Neuroprosthesis Device - Upper Extremity (NP-UE) in individuals living with cervical SCI.

DETAILED DESCRIPTION:
The Networked Neuroprosthesis(NNP) is an implantable, configurable neuromodulation platform that provides functional movement by the coordinated activation of peripheral neural pathways activating innervated paralyzed muscles, and sensing of physiological signals. The NNP-UE Configuration activates nerves of the upper extremity (arm and hand), and senses voluntary motion and/or electromyogram (EMG) in order to provide hand grasp.

The proposed work is focused on restoration of hand and reaching functions for people with cervical level spinal cord injury. For individuals who have sustained this injury, restoration of hand function is their top priority, and existing alternatives are limited. Neuroprosthesis are the most promising method for significant gain in hand and arm function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age > 16 years.
* Cervical level spinal cord injury, as defined by:

  1. International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) motor level of C1 through C7 and
  2. American Spinal Injury Association (ASIA) Impairment Scale (AIS) grade A, B, or C;
* Six months or more post-injury (neurostability);
* Neurologically stable following any nerve transfers affecting the upper extremity (typically, one year post surgery);
* Musculoskeletally and neurologically stable following any tendon transfers affecting the upper extremity (typically, 6-months).
* Peripheral nerve innervation to upper extremity muscles, including a grade 3/5 or higher Stimulated Manual Muscle Test (SMMT) strength in at least two of the following muscles in one arm:

  1. Adductor Pollicus, Abductor Pollicus Brevis (AbPB), Flexor Pollicus Longus (FPL), Extensor Pollicus Longus (EPL)/Extensor Pollicus Brevis (EPB), Extensor Digitorum Communis (EDC), Flexor Digitorum Superficialis (FDS), Flexor Digitorum Profundus (FDP), Pronator Quadratus (PQ), Extensor Carpi Ulnaris (ECU), Extensor Carpi Radialis Brevis (ECRB), Extensor Carpi Radialis Longus (ECRL), Flexor Carpi Ulnaris (FCU), Flexor Carpi Radialis (FCR), First Dorsal Interosseous(1DI), triceps,
  2. At least two of the grade 3/5 or higher excitable muscles must also have grade 2/5 or lower voluntary strength;
* Good proximal upper extremity strength as defined by biceps/brachialis/brachioradialis strength of 2/5 or higher on Manual Muscle Test on the side intended for implantation;
* Medically stable;
* Able to understand and provide informed consent.

Exclusion Criteria:

* Other neurological conditions (MS(multiple Sclerosis), diabetes with peripheral nerve involvement); Associated peripheral nerve / brachial plexus injury
* Progressive SCI;
* Co-existing cervical spine pathology (syrinx, unstable segment)
* Active implantable medical device (AIMD) such as a pacemaker or defibrillator;
* Active untreated infection such as pressure injury, urinary tract infection, pneumonia;
* History of coagulopathy, HIV, cardiopulmonary disease, bradycardia, poorly controlled autonomic dysreflexia, or chronic obstructive pulmonary disease that would preclude safe participation in the trial as determined by the investigator;
* Unhealed fractures that prevent functional use of arm;
* Extensive upper extremity denervation (fewer than two excitable hand muscles);
* Involvement in other ongoing clinical studies that exclude concurrent involvement in this study;
* Disorder or condition that requires MRI monitoring;
* Mechanical ventilator dependency;
* Currently pregnant (neuroprosthesis implantation delayed until no longer pregnant);
* Presence of disease that might interfere with participant safety, compliance, or evaluation of the condition under study;
* Other significant medical findings that, in the opinion of the investigator, preclude safe participation in the trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2022-01-23 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Grasp-Release Test | Pre-implant and three months post-implant, 6 months post implant, 12 months post implant
  Ability to pick up, move, and release six standard objects

SECONDARY OUTCOMES:
Change in Grasp Dynameter(force) | Pre-implant and three months post-implant, 6 months post implant, 12 months post implant
  Measure of muscular strength or the maximum force/tension generated by one's forearm muscles.
Change in Canadian Occupational Performance Measure (COPM) | Pre-implant and three months post-implant, 6 months post implant, 12 months post implant
  Evidence-based outcome measure designed to capture a client's self-perception of performance in everyday living, over time
Change in Activities of Daily Living (ADL) Abilities Test | Pre-implant and three months post-implant, 6 months post implant, 12 months post implant
  The Activities of Daily Living (ADL) profile uses both observation and interview to assess function in tasks completed in the personal, home, and community environments.
Change in Spinal Cord Independence Measure III (SCIM-III) | Pre-implant and three months post-implant, 6 months post implant, 12 months post implant
  The measure address three specific areas of function in patients with spinal cord injuries (SCI). It looks at self-care (feeding, grooming, bathing, and dressing), respiration and sphincter management, and a patient's mobility abilities (bed and transfers and indoors/outdoors)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Bryden, PhD, OTR/L, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ho CH, Triolo RJ, Elias AL, Kilgore KL, DiMarco AF, Bogie K, Vette AH, Audu ML, Kobetic R, Chang SR, Chan KM, Dukelow S, Bourbeau DJ, Brose SW, Gustafson KJ, Kiss ZH, Mushahwar VK. Functional electrical stimulation and spinal cord injury. Phys Med Rehabil Clin N Am. 2014 Aug;25(3):631-54, ix. doi: 10.1016/j.pmr.2014.05.001. PMID 25064792
- [Background] Peckham PH, Kilgore KL. Challenges and opportunities in restoring function after paralysis. IEEE Trans Biomed Eng. 2013 Mar;60(3):602-9. doi: 10.1109/TBME.2013.2245128. Epub 2013 Mar 7. PMID 23481680
- [Background] Makowski N, Campean A, Lambrecht J, Buckett J, Coburn J, Hart R, Miller M, Montague F, Crish T, Fu M, Kilgore K, Peckham PH, Smith B. Design and Testing of Stimulation and Myoelectric Recording Modules in an Implanted Distributed Neuroprosthetic System. IEEE Trans Biomed Circuits Syst. 2021 Apr;15(2):281-293. doi: 10.1109/TBCAS.2021.3066838. Epub 2021 May 25. PMID 33729949
- See also: Cleveland Functional Electrical Stimulation Center — https://fescenter.org/